CLINICAL TRIAL: NCT02234375
Title: Efficacy of Gadolinium Contrast in CT Pulmonary Angiography in Patients With Allergy to Iodine
Brief Title: Use of Gadolinium in CT Pulmonary Angiography
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Gadolinium attenuation in vitro inadequate
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amita Sharma, MD, Radiologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012P002535b
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; Contrast; Computed tomography; Gadolinium
MeSH Terms: conditions — Pulmonary Embolism | interventions — Gadolinium; gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gadolinium enhancement (Experimental): Gadolinium enhancement will be performed using intravenous Dotarem[recommended dose of 0.2 mL/kg (0.1 mmol Gd/kg )]
  Interventions: Drug: Gadolinium

INTERVENTIONS:
Drug: Gadolinium — agents will be administered intravenously and a CT scan will be performed to evaluate contrast enhancement characteristics of the agents to assess their feasibility as an alternative to Iodine based contrast agents
  Other Names: Dotarem

SUMMARY:
The study will investigate patients with clinical suspicion for pulmonary embolism (PE) who have a contraindication to iodine based contrast. These patients normally get investigated with studies such as ultrasound and nuclear medicine studies but the fastest and preferred investigation is CT with contrast to look for filling defects in the pulmonary arteries. The investigators will assess whether gadolinium, which is currently used with MRI can be used with CT as an alternative effective contrast in diagnosis or exclusion of PE. A new type of CT scanner, a Dual Energy Scanner will be used to improve the visibility of Gadolinium contrast on CT.

DETAILED DESCRIPTION:
Contrast enhancement with Gadolinium will be evaluated to assess its efficacy for diagnosis and exclusion of pulmonary embolism in a patient who previously would not have been investigated with CTPA due to an underlying allergy to contrast or other contraindication. If this proves beneficial, it will allow such patients to be investigated successfully with CTPA

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of having a Pulmonary embolus
* Allergy to Iodine based intravenous contrast

Exclusion Criteria:

* Renal impairment
* Less than 20 years of age
* Non-English speaking
* Pregnancy
* Allergy to Gadolinium

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Pulmonary Embolism | 24 hours
  Ability of Gadolinium to diagnose pulmonary embolism on a dual energy CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States